CLINICAL TRIAL: NCT04679246
Title: Participatory Intervention to Improve Nutrition and Physical Activity in Schoolchildren From Acatlán de Juárez, Jalisco
Acronym: Acatlan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iberoamerican Institute of Sports Science and Human Movement (Other)
Collaborators: University of Guadalajara (Other); Mexican National Institute of Public Health (Other Government); Instituto Tecnológico y de Estudios Superiores de Occidente (Other)
Responsible Party: Principal Investigator, Cesar Octavio Ramos Garcia, PhD, Head of Research and Development, Iberoamerican Institute of Sports Science and Human Movement
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IICDEM-ID-001-2015
Record Dates: First submitted 2020-08-28; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Sedentary Behavior; Adipose Tissue; Child Obesity
Keywords: Child Obesity; Exercise; Healthy Eating; Anthropometry
MeSH Terms: conditions — Sedentary Behavior; Pediatric Obesity; Motor Activity | interventions — Diet, Healthy; Exercise

STUDY DESIGN:
Intervention Model Description: Monitoring and evaluation of the impact of the intervention will be carried out through a community trial. There will be three schools in each study group (intervention and control). There will be three measurement periods: a baseline in the 2015-2016 school year, an intermediate measurement in the 2016-2017 school year, and a final measurement in the 2017-2018 school year. The measurement periods will have an estimated duration of two months.
  In the measurement periods, the body composition of the children from 1st to 4th grade will be obtained, and they will be followed up for two years; The dynamics of water and food consumption, physical activity, functional physical capacities, as well as availability and accessibility of food in schools will be identified. In addition, from a sub-sample of the study subjects, questionnaires on the frequency of food consumption, additional anthropometric measurements, and venous blood will be obtained to determine glucose and blood lipid levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General Intervention (Experimental): The strategies will be implemented in the three intervention elementary schools. The schools were conveniently chosen for the size of the student population. In addition to having a sufficient population, it was important that the authorities of each school site agreed to participate.
  Interventions: Behavioral: Participatory intervention
- Subsample intervention (Experimental): A group will be randomly selected from each school grade from the intervention schools, and within each chosen group 12 children will be randomly selected per group (48 children in total per school).
  Interventions: Behavioral: Participatory intervention
- Control (No Intervention): Three primary schools were selected from a close locality (Villa Corona, Jalisco). This was chosen because it is similar in relation to the social, economic, and geographical context to the locality of intervention. The schools were selected for the similarity in the size of the student population of the intervention schools.

INTERVENTIONS:
Behavioral: Participatory intervention — Surveillance in compliance with the regulation of the sale of food in school buildings, according to official guidelines Training for the preparation of hygienic and healthy food for the personnel in charge of food sale Promotion of the consumption of simple water and healthy foods Reconditioning of the infrastructure for the consumption of simple water, free and healthy food, and the realization of physical activity Organization of events and support in the coordination of groups that promote physical activity at the community level Optimization of physical education classes at school sites Implementation of health promotion and care actions in the school context Development of skills in the school community for health care and generation of healthy school environments Creation and strengthening of health and nutrition committees in schools, with the participation of directors, teachers and parents to generate necessary and permanent conditions that favor healthy environments
  Other Names: Healthy diet; Physical activity; Nutrition literacy
  Arms: General Intervention; Subsample intervention

SUMMARY:
This is a community project carried out jointly by the Technological Institute of Higher Studies of the West (ITESO), the University Center of Tonalá of the University of Guadalajara (CUTonalá) and the University Center of Health Sciences of the University of Guadalajara ( CUCS) with advice from the National Institute of Public Health (INSP), financed by the Tresmontes Lucchetti company and endorsed by the Jalisco Association of Nutritionists, AC (AJANUT). This project follows the provisions of the "National Strategy for the Prevention and Control of Overweight, Obesity and Diabetes" signed by the executive branch of the Federal Government. In particular, this project is inserted within the Public Health Strategy, in the strategic axis of Health Promotion and educational communication (while still having an impact on the axes of Epidemiological Surveillance and Prevention). In addition, it follows the agreement in which the general guidelines for the expenditure and distribution of food and beverages prepared and processed in the schools of the National Educational System were obtained, proposed by the Ministries of Health and Public Education. The aforementioned referrals are intended to protect and improve the health of Mexican children.

DETAILED DESCRIPTION:
The project is a community trial that will last three years, which includes an intervention group and a control group of three schools each. Acatlán de Juárez has a total of 11 elementary schools.

The strategies will be implemented in collaboration with the authorities of the Acatlán de Juárez community, the school authorities, ITESO staff, CUTonalá, CUCS, and AJANUT. Key actors from both the school and community levels will be involved through the study to adapt the strategies socially and culturally to promote community project ownership. An initial study of the viability of the project and the current conditions of food and physical activity in school facilities will be carried out, as well as the perception of the community. The research team will design the contents and materials of the intervention taking into account the opinions and suggestions of the community and the results of the initial study. The schools of the control group will be chosen from the municipality of Villa Corona, Jalisco, which is similar to Acatlán de Juárez.

The strategies proposed for intervention by the research team, which will be agreed with the community, including the following:

* Surveillance in compliance with the regulation of the sale of food in school buildings, according to official guidelines
* Sensitization of children, parents, teachers (especially those in charge of the physical education class) and personnel in charge of the food supply (school cooperative), to improve acceptance and commitment to the regulation of the sale of food
* Training for the preparation of hygienic and healthy food for the personnel in charge of food sale
* Promotion of the consumption of simple water and healthy foods
* Rescue and promotion of the consumption of regional foods
* Reconditioning of the infrastructure for the consumption of simple water, free and healthy food, and the realization of physical activity
* Organization of events and support in the coordination of groups that promote physical activity at the community level
* Optimization of physical education classes at school sites
* Implementation of health promotion and care actions in the school context
* Development of skills in the school community for health care and generation of healthy school environments
* Creation and strengthening of health and nutrition committees in schools, with the participation of directors, teachers and parents to generate necessary and permanent conditions that favor healthy environments

To achieve a greater rapprochement with the population, qualitative instruments will also be implemented before the intervention, such as focus groups and in-depth interviews, which allow the identification of barriers and possible solutions to improve eating habits and promote physical activity in the population. Likewise, during the intermediate and final measurement phases, similar qualitative strategies will be applied to rescue successes and points for improvement of the intervention.

During the implementation of the strategies, meticulous monitoring of the localities will be carried out to identify significant changes that may affect the eating habits and physical activity in either of the two groups (intervention and control).

ELIGIBILITY:
Inclusion Criteria:

* Children 6 to 10 years of age (completed at the beginning of the study) attending public schools.
* Mothers and fathers of school-age children.
* Responsible for cooperatives and school canteens.
* Key actors and members of the different groups involved in the implementation of the strategies.

Exclusion Criteria:

* Chronic disease with a confirmed diagnosis (cancer, type 1 or type 2 diabetes).
* Physical limitations that could affect development and normal eating patterns.
* Use of medications that can influence energy consumption and expenditure (for example, antidepressant drugs, antipsychotics, steroids).
* Children who are or were in a weight reduction program in the last year.
* Use of medications or confirmed diagnosis of diseases that could alter laboratory values.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Child overweigth and obesity | 3 years
  Shift prevalence of children overweigth and obesity

SECONDARY OUTCOMES:
Daily stepcount | 3 years
  Change childrens daily average stepcount
Physical fitness score | 3 years
  Change childrens physical fitness score measured by EUROFIT protocol
Self-efficacy | 3 years
  Change in children's perceptions about their capability to change their eating behavior. (A self-administered validated questionnaire, Likert scale, points summary obtained)
Attitudes | 3 years
  Change in negative or positive perceptions about target eating behaviors. (A self-administered validated questionnaire, Likert scale, points summary obtained)
Intention to change | 3 years
  Change in short term intentions to adopt a desirable eating behavior. (A self-administered validated questionnaire, Likert scale, points summary obtained)
Fruit and vegetable intake during school recess | 3 years
  Change in fruit and vegetable intake (g) during school recess. (Direct observation and weighted foods)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Patricia Arellano Gomez, PhD, Principal Investigator — Instituto Tecnologico y de Estudios Superiores de Occidente; Clio Chavez Palencia, PhD, Principal Investigator — University of Guadalajara; Hector Ochoa Gonzalez, MSc, Study Director — Instituto Tecnologico y de Estudios Superiores de Occidente; Oscar Loreto Garibay, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Iberoamerican Institute of Sports Science and Human Movement, Zapopan, Jalisco, Mexico

REFERENCES:
- [Result] Valencia-Sosa E, Chavez-Palencia C, Romero-Velarde E, Larrosa-Haro A, Vasquez-Garibay EM, Ramos-Garcia CO. Neck circumference as an indicator of elevated central adiposity in children. Public Health Nutr. 2019 Jul;22(10):1755-1761. doi: 10.1017/S1368980019000454. Epub 2019 Apr 2. PMID 30935440
- [Result] Ramos García, C. O., Loreto Garibay, O., & Ochoa González, H. (2017). Diagnostic precision of the submandibular skinfold, minimum waist circumference and minimum waist to height ratio, as adipose overweight and obesity indicators in children. Nutricion Clinica y Dietetica Hospitalaria, 37(2). https://doi.org/10.12873/372cesarramos

DOCUMENTS (2):
  • Study Protocol (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04679246/Prot_000.pdf
  • Informed Consent Form (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04679246/ICF_001.pdf